CLINICAL TRIAL: NCT01272193
Title: A Trial Comparing Efficacy and Safety of Insulin Degludec/Insulin Aspart With Insulin Glargine in Insulin Naive Subjects With Type 2 Diabetes (BOOST™: JAPAN)
Brief Title: Comparison of NN5401 With Insulin Glargine in Insulin Naive Subjects With Type 2 Diabetes
Acronym: BOOST™
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN5401-3896; U1111-1118-0124 (Other: WHO); JapicCTI-111385 (Registry Identifier: JAPIC)
Record Dates: First submitted 2011-01-06; First posted 2011-01-07 (Estimated); Results first posted 2015-11-23 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin degludec, insulin aspart drug combination; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDegAsp OD (Experimental)
  Interventions: Drug: insulin degludec/insulin aspart; Drug: insulin glargine
- IGlar OD (Active Comparator)
  Interventions: Drug: insulin glargine

INTERVENTIONS:
Drug: insulin degludec/insulin aspart — Injected subcutaneously (under the skin) once daily prior to the largest meal of the day as monotherapy or combined with no more than 2 oral anti-diabetic drugs (OADs).
  Arms: IDegAsp OD
Drug: insulin glargine — Administered according to approved labelling either as monotherapy or combined with no more than 2 OADs.

SUMMARY:
This trial is conducted in Japan. The aim of this trial is to investigate the efficacy and safety of NN5401 (insulin degludec/insulin aspart) with insulin glargine in subjects with type 2 diabetes in Japan. Depending on pre-trial oral anti-diabetic drugs (OADs), subjects continued at the same dose and dosing frequency.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus (diagnosed clinically) for at least 6 months
* HbA1c 7.0-10.0% (both inclusive) by central laboratory analysis
* Body Mass Index (BMI) below or equal to 35.0 kg/m^2
* Insulin naive subject and ongoing treatment with 1 or more oral antidiabetic drugs (OADs) for at least 12 weeks prior to randomisation with at least recommended maintenance dose according to local, approved labelling Allowed are: a. Previous short term insulin treatment up to 14 days; b. Treatment during hospitalization or during gestational diabetes is allowed for periods longer than 14 days)

Exclusion Criteria:

* Anticipated change in concomitant medication known to interfere significantly with glucose metabolism, such as systemic corticosteroids, beta-blockers, mono amino oxidase (MAO) inhibitors
* Use of glucagon-like peptide-1 (GLP-1) receptor agonists, buformine and/or rosiglitazone within the last 12 weeks prior to randomisation
* Cardiovascular disease, within the last 6 months prior to Visit 1, defined as: stroke; decompensated heart failure New York Heart Association (NYHA) class III or IV; myocardial infarction; unstable angina pectoris; or coronary arterial bypass graft or angioplasty

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2011-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (45):
- Japan (45):
  - Novo Nordisk Investigational Site, Asahikawa-shi, Hokkaido
  - Novo Nordisk Investigational Site, Chigasaki-shi, Kanagawa
  - Novo Nordisk Investigational Site, Chuo-ku, Tokyo
  - Novo Nordisk Investigational Site, Ebina-shi
  - Novo Nordisk Investigational Site, Fukuoka-shi, Fukuoka
  - Novo Nordisk Investigational Site, Iruma-shi, Saitama
  - Novo Nordisk Investigational Site, Izumisano
  - Novo Nordisk Investigational Site, Kamakura-shi
  - Novo Nordisk Investigational Site, Kanagawa-shi, Yokohama
  - Novo Nordisk Investigational Site, Kashiwa-shi, Chiba
  - Novo Nordisk Investigational Site, Kashiwara-shi, Osaka
  - Novo Nordisk Investigational Site, Katsushika-ku, Tokyo
  - Novo Nordisk Investigational Site, Kawagoe-shi, Saitama
  - Novo Nordisk Investigational Site, Kitakyushu-shi, Fukuoka
  - Novo Nordisk Investigational Site, Koriyama-shi, Fukushima
  - Novo Nordisk Investigational Site, Kumamoto-shi, Kumamoto
  - Novo Nordisk Investigational Site, Kumamoto-shi,Kumamoto
  - Novo Nordisk Investigational Site, Kurume-shi, Fukuoka
  - Novo Nordisk Investigational Site, Kyoto-shi, Kyoto
  - Novo Nordisk Investigational Site, Matsumoto-shi, Nagano
  - Novo Nordisk Investigational Site, Miyazaki
  - Novo Nordisk Investigational Site, Naha
  - Novo Nordisk Investigational Site, Naka-shi, Ibaraki
  - Novo Nordisk Investigational Site, Nishinomiya-shi, Hygo
  - Novo Nordisk Investigational Site, Obihiro-shi, Hokkaido
  - Novo Nordisk Investigational Site, Ogawa
  - Novo Nordisk Investigational Site, Okawa-shi, Fukuoka
  - Novo Nordisk Investigational Site, Ota-ku, Tokyo
  - Novo Nordisk Investigational Site, Oyama-shi, Tochigi
  - Novo Nordisk Investigational Site, Ōita
  - Novo Nordisk Investigational Site, Sapporo, Hokkaido
  - Novo Nordisk Investigational Site, Sapporo-shi, Hokkaido
  - Novo Nordisk Investigational Site, Sappro-shi, Hokkaido
  - Novo Nordisk Investigational Site, Sasebo-shi, Nagasaki
  - Novo Nordisk Investigational Site, Sendai
  - Novo Nordisk Investigational Site, Shimotsuke-shi, Tochigi
  - Novo Nordisk Investigational Site, Shizuoka
  - Novo Nordisk Investigational Site, Tagajō-shi
  - Novo Nordisk Investigational Site, Tagawa-shi, Fukuoka
  - Novo Nordisk Investigational Site, Takatsuki-shi, Osaka
  - Novo Nordisk Investigational Site, Tamana-shi, Kumamoto
  - Novo Nordisk Investigational Site, Tokyo
  - Novo Nordisk Investigational Site, Tsuchiura-shi, Ibaraki
  - Novo Nordisk Investigational Site, Urasoe-shi,
  - Novo Nordisk Investigational Site, Yokohama-shi, Kanagawa

REFERENCES:
- [Result] Onishi Y, Ono Y, Rabol R, Endahl L, Nakamura S. Superior glycaemic control with once-daily insulin degludec/insulin aspart versus insulin glargine in Japanese adults with type 2 diabetes inadequately controlled with oral drugs: a randomized, controlled phase 3 trial. Diabetes Obes Metab. 2013 Sep;15(9):826-32. doi: 10.1111/dom.12097. Epub 2013 Apr 5. PMID 23557077
- [Derived] Yang W, Akhtar S, Franek E, Haluzik M, Hirose T, Kalyanam B, Kar S, Wu T, Gogas Yavuz D, Unnikrishnan AG. Postprandial Glucose Excursions in Asian Versus Non-Asian Patients with Type 2 Diabetes: A Post Hoc Analysis of Baseline Data from Phase 3 Randomised Controlled Trials of IDegAsp. Diabetes Ther. 2022 Feb;13(2):311-323. doi: 10.1007/s13300-021-01196-7. Epub 2022 Jan 19. PMID 35044568
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 48 sites in Japan.
Pre-assignment Details: Subjects continued on not more than 2 oral antidiabetic drugs (excluding sulphonylureas/dipeptyl peptidase-4 [DPP-4] inhibitors/glinides) at the pre-randomisation dose level and dosing frequency.
Groups:
- IDegAsp OD: Insulin degludec/insulin aspart (IDegAsp) was given subcutaneously once daily (OD) either as monotherapy or in combination with no more than 2 oral antidiabetic drugs (excluding sulphonylureas/DPP-4 inhibitors/glinides). IDegAsp was given just prior to the largest meal of the day. Insulin doses were individually adjusted.
- IGlar OD: Insulin glargine (IGlar) was given once daily (OD) according to approved labelling either as monotherapy or in combination with no more than 2 oral antidiabetic drugs (excluding sulphonylureas/DPP-4 inhibitors/glinides). IGlar was given before breakfast or at bedtime but at the same time each day. Insulin doses were individually adjusted.
Period: Overall Study
Arm/Group | IDegAsp OD | IGlar OD
Started | 147 | 149
Completed | 137 | 137
Not Completed | 10 | 12
Not completed — Adverse Event | 1 | 1
Not completed — Lack of Efficacy | 0 | 3
Not completed — Withdrawal Criteria | 1 | 1
Not completed — Unclassified | 8 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IDegAsp OD | IGlar OD | Total
Number analyzed (Participants) | 147 | 149 | 296
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (10.0) | 61.0 (9.6) | 60.5 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 50 | 107
  Male | 90 | 99 | 189
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 8.3 (0.8) | 8.5 (0.8) | 8.4 (0.8)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] | 9.0 (1.6) | 9.1 (1.9) | 9.0 (1.7)
Body weight [Mean (Standard Deviation); unit: kg] | 66.2 (13.4) | 66.4 (13.3) | 66.3 (13.4)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Haemoglobin (HbA1c)
Description: Observed change from baseline in HbA1c after 26 weeks of treatment
Time Frame: Week 0, Week 26
Population: Full analysis set (FAS) included all randomised subjects and missing data were imputed using last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | IDegAsp OD | IGlar OD
Number analyzed (Participants) | 147 | 149
percentage of glycosylated haemoglobin | -1.35 (0.86) | -1.22 (0.98)

2. Secondary Outcome: Mean Increment of 9-point Self Measured Plasma Glucose Profile (SMPG) at the Main Evening Meal
Description: Observed mean increment of the 9-point self-measured plasma glucose profile (SMPG) at the main evening meal
Time Frame: Week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDegAsp OD | IGlar OD
Number analyzed (Participants) | 147 | 149
mmol/L | 1.4 (4.2) | 4.7 (3.6)

3. Secondary Outcome: Rate of Treatment Emergent Adverse Events (AEs)
Description: Corresponds to rate of AEs per 100 patient years of exposure. Severity assessed by investigator. Mild: no or transient symptoms, no interference with subject's daily activities. Moderate: marked symptoms, moderate interference with subject's daily activities. Severe: considerable interference with subject's daily activities, unacceptable. Serious AE: AE that at any dose results in any of the following: death, a life-threatening experience, in-subject hospitalization/prolongation of existing hospitalisation, persistent/significant disability/incapacity/congenital anomaly/birth defect.
Time Frame: Week 0 to Week 26 + 7 days follow up
Population: Safety analysis set includes all subjects who received at least one dose of the investigational product or its comparator.
Measure: Number; unit: Events/100 years of patient exposure
Arm/Group | IDegAsp OD | IGlar OD
Number analyzed (Participants) | 147 | 149
Events/100 years of patient exposure
  Adverse events (AEs) | 334 | 368
  Serious AEs | 7 | 4
  Severe AEs | 1 | 0
  Moderate AEs | 17 | 14
  Mild AEs | 316 | 353
  Fatal AEs | 0 | 0

4. Secondary Outcome: Rate of Confirmed Hypoglycaemic Episodes
Description: Observed rate of confirmed hypoglycaemic episodes per 100 patient years of exposure (PYE). Confirmed hypoglycaemic episodes consisted of severe hypoglycaemia as well as minor hypoglycaemic episodes. Severe hypoglycaemic episodes were defined as requiring assistance to administer carbohydrate, glucagon, or other resuscitative actions. Minor hypoglycaemic episodes were defined as able to treat her/himself and plasma glucose below 3.1 mmol/L.
Time Frame: Week 0 to Week 26 + 7 days follow up
Population: as for outcome 3
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | IDegAsp OD | IGlar OD
Number analyzed (Participants) | 147 | 149
Episodes/100 years of patient exposure | 191 | 271

5. Secondary Outcome: Rate of Nocturnal Confirmed Hypoglycaemic Episodes
Description: Observed rate of confirmed hypoglycaemic episodes per 100 patient years of exposure (PYE). Confirmed hypoglycaemic episodes consisted of severe hypoglycaemia as well as minor hypoglycaemic episodes. Severe hypoglycaemic episodes were defined as requiring assistance to administer carbohydrate, glucagon, or other resuscitative actions. Minor hypoglycaemic episodes were defined as able to treat her/himself and plasma glucose below 3.1 mmol/L. Nocturnal hypoglycaemic episodes were defined as occurring between 00:01 and 05:59 a.m.
Time Frame: Week 0 to Week 26 + 7 days follow up
Population: Safety analysis set included all subjects who received at least one dose of the investigational product or its comparator.
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | IDegAsp OD | IGlar OD
Number analyzed (Participants) | 147 | 149
Episodes/100 years of patient exposure | 39 | 53

6. Secondary Outcome: Change in Body Weight
Description: Observed change from baseline in body weight after 26 weeks of treatment
Time Frame: Week 0, Week 26
Population: Safety analysis set includes all subjects who received at least one dose of the investigational product or its comparator. Missing data is imputed using last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | IDegAsp OD | IGlar OD
Number analyzed (Participants) | 147 | 149
kg | 0.7 (2.8) | 0.7 (2.2)

ADVERSE EVENTS:
Time Frame: The adverse events were collected in a time frame of 26 weeks + 7 days follow up.
Description: Safety analysis set includes all subjects who received at least one dose of the investigational product or its comparator.
Arm/Group | IDegAsp OD | IGlar OD
Serious Adverse Events (participants affected / at risk) | 5/147 | 3/149
Other Adverse Events (participants affected / at risk) | 37/147 | 47/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDegAsp OD (N=147) | IGlar OD (N=149)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Osteitis condensans (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDegAsp OD (N=147) | IGlar OD (N=149)
Diabetic retinopathy (Eye disorders) | 8 (9) | 10 (10)
Nasopharyngitis (Infections and infestations) | 33 (39) | 38 (45)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.